CLINICAL TRIAL: NCT05032040
Title: A Phase 2 Study of XmAb20717 in Patients With Selected Gynecological Malignancies and Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of XmAb20717 (Vudalimab)in Patients With Selected Advanced Gynecologic and Genitourinary Malignancies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XmAb20717-05
Record Dates: First submitted 2021-08-31; First posted 2021-09-02 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer; Clear Cell Carcinoma; Endometrial Cancer; Cervical Carcinoma; Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Keywords: Endometrial Cancer; Ovarian Cancer; Cervical Cancer; Prostate Cancer; Gynecological Cancer,; Fallopian Tube Cancer; Peritoneal Cancer; Clear Cell Carcinoma; vudalimab; XmAb20717
MeSH Terms: conditions — Ovarian Neoplasms; Adenocarcinoma, Clear Cell; Endometrial Neoplasms; Uterine Cervical Neoplasms; Prostatic Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- vudalimab (Experimental)
  Interventions: Biological: vudalimab

INTERVENTIONS:
Biological: vudalimab — Monoclonal bispecific antibody

SUMMARY:
This is a Phase 2, multicenter, two-stage, open-label, parallel-group study designed to evaluate the efficacy and safety of vudalimab (XmAb20717) in patients with selected advanced gynecologic and genitourinary malignancies.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, two-stage, open-label, parallel-group study designed to evaluate the efficacy and safety of vudalimab in patients with selected advanced gynecologic and genitourinary malignancies and to identify tumor types for further evaluation.

In Stage 1, subjects will be enrolled into 1 of 5 tumor-specific, parallel cohorts (n = 10 each):

* Platinum-resistant high-grade serous ovarian cancer (HGSOC)
* Chemotherapy relapsed or refractory clear cell ovarian, endometrial, or peritoneal cancer
* Immune-checkpoint-inhibitor-refractory microsatellite stable (MSS) endometrial cancer (EC)
* Previously treated recurrent or metastatic cervical cancer
* Metastatic castration-resistant prostate cancer (mCRPC)

Within each tumor-specific cohort in Stage 1, a primary endpoint of ORR at 12 weeks, based on Investigator review, will be used to determine cohort expansion into Stage 2. Each Stage 1 cohort that achieves an ORR of ≥ 20% (at least 2 out of 10 subjects with an objective response) will enroll up to an additional 20 subjects in Stage 2. Cohorts with an ORR of less than 20% will discontinue enrollment. However, additional factors will be considered in determining an expansion into Stage 2 (eg, enrollment rate, complete versus partial response, and duration of response [DOR].

In Stage 2, up to 20 additional subjects with mCRPC with or without measurable disease will be enrolled; the primary endpoint is PSA50.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Adult (age ≥ 18 years)
* Cancer must have progressed after treatment with standard of care therapy approved for the treatment of that indication
* Histologically confirmed diagnosis of one of the following tumor types, along with clinical/pathologic confirmation of the additional requirements for each indication, as appropriate:

  1. Persistent or recurrent clear cell carcinoma of the ovary, peritoneum, or endometrium after treatment with platinum-based systemic chemotherapy
  2. Persistent or recurrent high-grade serous carcinoma of the ovary, fallopian tube, or peritoneum after treatment with platinum-based systemic chemotherapy (except subjects with a diagnosis of carcinosarcoma)
  3. Recurrent or metastatic cervical carcinoma previously treated with standard-of-care systemic chemotherapy and FDA-approved immunotherapy, if eligible
  4. Advanced endometrial carcinoma that is not microsatellite instability-high (MSI-H) or deficient mismatch repair (dMMR) in patients who are not candidates for curative surgery or radiation, and that has progressed following treatment with no more than one prior line of systemic therapy and prior treatment with FDA-approved combination therapy consisting of a checkpoint inhibitor and a targeted agent
  5. For patients with mCRPC castration-resistant prostate cancer defined as progressive disease (PD) after surgical castration, or progression in the setting of medical androgen ablation with a castrate level of testosterone (< 50 ng/dL)
  6. Documented progressive mCRPC based on at least 1 of the following:
* PSA progression, defined as at least 2 rises in PSA with a minimum of a 1-week interval
* Soft-tissue progression per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Progression of bone disease (evaluable disease) or 2 or more new bone lesions by bone scan
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) in Stage 1
* Patients with mCRPC without measurable disease are eligible in for Stage 2
* Adequate available archival formalin-fixed paraffin-embedded block(s)/slides containing tumor and/or adequate predose fresh tumor biopsy tissue
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Female subjects of childbearing potential must agree to use a highly effective method of birth control during and for 4 weeks after the last dose of XmAb20717. Women are considered to be of childbearing potential unless it is documented that they are over the age of 60 OR postmenopausal by history with no menses for 1 year and confirmed by follicle-stimulating hormone (using local reference ranges) OR have a history of hysterectomy and/or bilateral oophorectomy OR have a history of bilateral tubal ligation.
* Fertile male subjects must be willing to practice a highly effective method of birth control during and for 4 weeks after last dose of XmAb20717
* Male subjects must agree not to donate sperm from screening through 4 weeks after last dose of XmAb20717
* Able and willing to complete the entire study according to the study schedule

Exclusion Criteria:

* Subjects currently receiving other anticancer therapies, except that subjects with mCRPC may continue to receive luteinizing hormone-releasing hormone (LHRH) analogue therapy
* More than 2 prior chemotherapy regimens for subjects in the cervical cancer, CCC, HGSOC, or mCRPC cohorts
* Progression on more than 2 prior lines of androgen receptor signal inhibitor therapy (mCRPC cohort)
* Prior treatment with a CTLA4-targeted agent
* Prior treatment with nivolumab, pembrolizumab, or any other PD1-, PDL1- or programmed cell death ligand 2- (PDL2)-directed therapy, except that:

  1. Subjects with MSS EC may have received anti-PD1 therapy as part of an FDA-approved regimen in the approved disease setting
  2. Subjects with cervical cancer may have received anti-PD1 therapy as an FDA-approved agent in an approved disease setting
* Treatment with any other anticancer therapy within 2 weeks of the start of study drug (ie, other immunotherapy, chemotherapy, radiation therapy, etc.)
* A life-threatening (Grade 4) immune-mediated adverse event (AE) associated with prior administration of an immunotherapy agent
* Failure to recover from any immunotherapy-related toxicity from prior cancer therapy to ≤ Grade 1, except that subjects are eligible if a previous immunotherapy-related endocrinopathy is medically managed with hormone replacement therapy only
* Failure to recover from any other cancer therapy-related toxicity (other than immune-related toxicity) related to previous anticancer treatment to ≤ Grade 2
* Have known active central nervous system metastases and/or carcinomatous meningitis
* Platelet count < 100 × 109/L
* Hemoglobin level ≤ 9.0 g/dL
* Absolute neutrophil count < 1.5 × 109/L
* Aspartate aminotransferase (AST) at screening > 3 × upper limit of normal (ULN) for subjects without known liver involvement by tumor; or > 5 × ULN for subjects with known liver involvement by tumor
* Alanine aminotransferase (ALT) at screening > 3 × ULN for subjects without known liver involvement by tumor; or > 5 × ULN for subjects with known liver involvement by tumor
* Bilirubin ≥ 1.5 × ULN (unless prior diagnosis and documentation of ongoing hemolysis or Gilbert's syndrome has been made)
* Estimated creatinine clearance < 50 mL/minute calculated by the Cockcroft Gault or Modification of Diet in Renal Disease formulas
* Active known or suspected autoimmune disease (except that subjects are permitted to enroll if they have vitiligo; type 1 diabetes mellitus or residual hypothyroidism due to an autoimmune condition that is treatable with hormone replacement therapy only; autoimmune adrenal insufficiency that is managed with low-dose corticosteroids; psoriasis, atopic dermatitis, or another autoimmune skin condition that is managed without systemic therapy; or arthritis that is managed without systemic therapy beyond oral acetaminophen and nonsteroidal anti-inflammatory drugs)
* • Has any condition requiring systemic treatment with corticosteroids, prednisone equivalents, or other immunosuppressive medications within 14 days prior to first dose of XmAb20717 (except that inhaled or topical corticosteroids or brief courses of corticosteroids given for prophylaxis of contrast dye allergic response are permitted)
* Receipt of an organ allograft
* History of small or large bowel obstruction within 3 months of enrollment, including subjects with palliative gastric drainage catheters. Subjects with palliative diverting ileostomy or colostomy are allowed if they have been symptom-free for more than 3 months.
* Ongoing bowel perforation or presence of bowel fistula or intra-abdominal abscess
* Subjects with refractory ascites, for example, ascites needing drainage catheter or therapeutic paracentesis more often than every 4 weeks
* Histologic diagnosis of carcinosarcoma of the ovary
* Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression
* History or evidence of any other clinically unstable/uncontrolled disorder, condition, or disease (including, but not limited to, cardiopulmonary, renal, metabolic, hematologic, or psychiatric) other than their primary malignancy, that, in the opinion of the Investigator, would pose a risk to patient safety or interfere with study evaluations, procedures, or completion
* Evidence of any serious bacterial, viral, parasitic, or systemic fungal infections within the 30 days prior to the first dose of study drug
* Receipt of a live-virus vaccine within 30 days prior to first dose of study drug (Seasonal flu and COVID-19 vaccines are permitted, as long as they do not contain live virus. Seasonal flu vaccines should no be administered within 24 hours of planned administration of XmAb20717. COVID-19 vaccines should be administered 48 to 72 hours before or after XmAb20717 dosing
* Known HIV-positive subject with CD4+ T-cell (CD4+) counts < 350 cells/μL, or an HIV viral load greater than 400 copies/mL, or a history of an AIDS-defining opportunistic infection within the past 12 months, or who has not been on established antiretroviral therapy (ART) for at least 4 weeks prior to initiation of XmAb20717 dosing. (Effective ART is defined as a drug, dosage, and schedule associated with reduction and control of the viral load. HIV positive subjects who do not meet any of these exclusion criteria are eligible.)
* Positive test for hepatitis C RNA (a subject who is hepatitis C virus [HCV] antibody positive but HCV RNA negative due to documented, curative prior antiviral treatment or natural resolution is eligible)
* Positive test for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb); a subject whose HBsAg is negative and HBcAb is positive may be enrolled if a hepatitis B virus (HBV) DNA test is negative and the subject is retested for HBsAg and HBV DNA every 2 months.
* Subject is pregnant or breastfeeding or planning to become pregnant while enrolled in the study, up to the final end-of-treatment visit
* Positive urine pregnancy test (ie, urine human chorionic gonadotropin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
PSA50 is the primary endpoint for the mCRPC cohort. Objective Response Rate (ORR) as assessed by Response Evaluation Criteria in Solid Tumours (RECIST) version 1 criteria is the primary endpoint for gynecological malignancy cohorts | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jolene Shorr, Study Director — Xencor, Inc.
Locations (17):
- United States (17):
  - Arizona Oncology Associates, PC - NAHOA, Prescott, Arizona
  - UCSD Moores Cancer Center, La Jolla, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Kaiser Permanente Medical Group, Riverside, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada-Southern Hills, Las Vegas, Nevada
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Texas Oncology - Central South, Austin, Texas
  - Virginia Oncology Associates, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No